CLINICAL TRIAL: NCT03842670
Title: Neurocognitive and Neurobehavioral Mechanisms of Change Following Psychological
Brief Title: Neurocognitive and Neurobehavioral Mechanisms of Change Following Psychological Treatment for Alcohol Use Disorder
Acronym: ABQTREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Barbara S McCrady, PhD, Distinguished Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1240557-4
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse; Alcohol Drinking; Alcohol Dependence
Keywords: Alcohol Use Disorder; Behavioral Treatment; Mechanisms of behavior change; Neuroimaging
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-Behavior Therapy (Active Comparator): The CBT condition will include 8 weekly, 60-minute sessions, and will be delivered according to the Epstein & McCrady (2009) cognitive-behavioral treatment manual, excluding material provided in the platform treatment. The treatment manual and accompanying client workbook provide detailed therapist instructions for each session, client exercises, worksheets, and homework assignments. The treatment focuses on cognitive and behavioral coping skills training, and emphasizes problem-solving as an overall approach to dealing with drinking.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Mindfulness Based Relapse Prevention (Active Comparator): The MBT condition will be adapted from the 8-week version of the mindfulness-based relapse prevention (MBRP) manual (Bowen et al., 2011; Witkiewitz et al., 2005). The main adaptation will be to eliminate the relapse prevention/CBT components and focus attention on mindfulness practices. The mindfulness practices in MBT are designed to increase awareness of triggers and decrease reactivity to distress or discomfort in the presence of triggers (Witkiewitz & Bowen, 2010). The relevant worksheets and homework assignments focusing on mindfulness tools will be maintained from the MBRP manual.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — The CBT condition will include 8 weekly, 60-minute sessions, and will be delivered according to the Epstein & McCrady (2009) cognitive-behavioral treatment manual, excluding material provided in the platform treatment. The treatment manual and accompanying client workbook provide detailed therapist instructions for each session, client exercises, worksheets, and homework assignments. The treatment focuses on cognitive and behavioral coping skills training, and emphasizes problem-solving as an overall approach to dealing with drinking. Treatment sessions may be audio-recorded for supervision and to ensure that the treatment is being delivered as intended.
  Arms: Cognitive-Behavior Therapy
Behavioral: Mindfulness Based Relapse Prevention — The MBT condition will be adapted from the 8-week version of the mindfulness-based relapse prevention (MBRP) manual (Bowen et al., 2011; Witkiewitz et al., 2005). The main adaptation will be to eliminate the relapse prevention/CBT components and focus attention on mindfulness practices. The mindfulness practices in MBT are designed to increase awareness of triggers and decrease reactivity to distress or discomfort in the presence of triggers (Witkiewitz & Bowen, 2010). The relevant worksheets and homework assignments focusing on mindfulness tools will be maintained from the MBRP manual. Treatment sessions may be audio-recorded for supervision and to ensure that the treatment is being delivered as intended.
  Arms: Mindfulness Based Relapse Prevention

SUMMARY:
Alcohol Use Disorder (AUD) is a significant public health problem, with prevalence rates of 13.9% for current and 29.1% for lifetime diagnosis (Grant et al., 2015). AUD creates harm at the individual, familial, and societal level, with an estimated societal cost of $249 billion (Sacks et al., 2015) per year. The course of AUD typically is characterized by periods of relapse to problematic drinking (Maisto et al., 2014), signaling a need for better treatments and understanding of mechanisms of behavior change.

The goal of this research is to conduct a randomized clinical trial with 140 participants who have an Alcohol Use Disorder (AUD). Each participant will complete behavioral assessments, self-report surveys and brain imaging before and after receiving psychotherapy treatment to change their drinking behaviors. Various aspects of behavior change will be looked at to better understand changes in brain function and emotional reactivity when someone changes their patterns of alcohol use. The two treatment used in this study have been found to be helpful in reducing alcohol use. Participants will be randomly assigned to either Mindfulness-Based Relapse Prevention (MBRP) or Cognitive Behavior Therapy (CBT) that will be completed in 12 weekly therapy sessions.

It is anticipated that there will be numerous changes in brain function that are found when someone reduces or stops their alcohol use after the completion of 12 weeks of treatment.

DETAILED DESCRIPTION:
Although pharmacological and psychosocial treatments for alcohol use disorders (AUDs) exist that improve outcomes over natural recovery (Finney et al., 2013), outcomes are still modest. Identifying mechanisms of behavior change (MOBCs) that lead to successful outcomes may be critical for efforts to improve existing treatments or to better match patients with particular treatments. The goal of the proposed research is to conduct a randomized clinical trial to systematically examine pretreatment neurocognitive and behavioral characteristics and changes in brain function over time during two empirically supported treatments for AUD. One hundred forty treatment-seeking individuals with an AUD will be randomized to receive either 8 weeks of Cognitive Behavioral Treatment (CBT) or Mindfulness Based Treatment (MBT) after receiving 4 weeks of a platform treatment that focuses on enhancing motivation to change. Neurocognitive and behavioral characteristics will be measured using neuroimaging, comprehensive behavioral assessments, and patient self-reports. To establish the temporal relationship between changes in drinking and changes in these MOBCs, patients will be assessed at: (a) baseline; (b) four weeks into treatment; (c) immediately post-treatment; and (d) 9- and 15-months post-baseline. Self-report measures and behavioral tasks will be administered at monthly intervals during treatment; and fMRI will be collected at baseline, and at 3, and 9-months post baseline. The primary aim of the study is to examine the effects of the treatments on three hypothesized mechanisms: craving/regulation of craving, cognitive and behavioral control, and regulation of affect/arousal. The secondary aim will identify neurocognitive and behavioral baseline characteristics predictive of reductions in drinking over time and differential patterns of response to CBT or MBT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-85 years
2. Self-identify as a heavy/binge/weekly drinker
3. Engage in "hazardous and harmful alcohol use" (Babor et al., 2001) based on an AUDIT score > 8 for men and > 7 for women
4. Breath alcohol level of 0.00 at in-person screening
5. Right handed
6. Explicitly be seeking help for their drinking
7. Alcohol use during the past 30 days

Exclusion Criteria:

1. History of brain injury or neurological diagnoses
2. Evidence of current psychosis
3. Past-year substance dependence other than nicotine or marijuana
4. Evidence of recent illicit drug (other than marijuana) use on a urine screen
5. Contraindications for MRI (e.g., medical devices in the body)
6. Female participants who think they may be pregnant must pass a urine pregnancy screen prior to each MRI scanning session
7. Estimated IQ < 80
8. Unable to read or speak English fluently
9. History of major alcohol withdrawal
10. Currently in treatment for alcohol use (or within the past 6 months)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Percent heavy drinking days | Baseline, 4-week within treatment visit, 8-week within treatment visit, and 3-month follow-up, 9-month follow-up, and 15-month follow-up
  The Form 90 will be used to derive estimates of the outcome: percent heavy drinking days, where heavy drinking is defined as 4+ drinks per occasion for women and 5+ drinks per occasion for men.

SECONDARY OUTCOMES:
Percent drinking days | Baseline, 4-week within treatment visit, 8-week within treatment visit, and 3-month follow-up, 9-month follow-up, and 15-month follow-up
  The Form 90 will be used to derive estimates of the outcome percent drinking days.
MOBC: Craving - self report | Up to 15 months
  The Penn Alcohol Craving Scale will be used to examine changes in craving that occur during and after treatment. Ratings range from 1-6, with higher scores indicating a higher level of craving.
MOBC: Regulation of Affect/Arousal - negative affect self-report | Up to 15 months
  The Negative Affect Summary score from the National Institutes of Health Negative Emotions toolbox will be used to assess overall negative affect changes during and after treatment. T-scores on the measure can range from 1-100, with higher scores indicating a higher level of negative affect.
MOBC: Regulation of Affect/Arousal - neuroimaging | Up to 9 months
  The difference in percent signal change during negative vs. neutral picture cues in amygdala will be assessed using a cue task while participants are scanned using functional magnetic resonance imaging.
MOBC: Cognitive and Behavioral Control - neuroimaging errors | Up to 9 months
  The difference in percent signal change during unsuccessful inhibition of responses vs. successful non-inhibition trials in dorsal anterior cingulate cortex will be assessed using a stop signal task while participants are scanned using functional magnetic resonance imaging.
MOBC: Cognitive and Behavioral Control - neuroimaging inhibition | Up to 9 months
  The difference in percent signal change during successful inhibition of responses vs. successful non-inhibition trials in right inferior frontal cortex will be assessed using a stop signal task while participants are scanned using functional magnetic resonance imaging.
MOBC: Cognitive and Behavioral Control - behavior | Up to 15 months
  The Monetary Choice Questionnaire will be used to determine the degree to which impulsive choice changes during and after treatment. A discounting rate (k) will be computed for each administration.
MOBC: Cognitive and Behavioral Control - self report impulsivity | Up to 15 months
  The UPPS-P Impulsive Behavior Scale will be used to examine changes in impulsivity that occur during and after treatment. Potential total scores range from 59-236, with higher scores indicating a higher level of impulsivity.
MOBC: Craving - neuroimaging | Up to 9 months
  The difference in percent signal change during alcohol vs. neutral picture cues in ventral striatum will be assessed using a cue task while participants are scanned using functional magnetic resonance imaging
Drinks per drinking day | Baseline, 4-week within treatment visit, 8-week within treatment visit, and 3-month follow-up, 9-month follow-up, and 15-month follow-up
  The Form 90 will be used to derive estimates of the outcome: drinks (standard drink=14 grams of pure alcohol) per drinking day.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara McCrady, PhD, Principal Investigator — The University of New Mexico
Locations (2):
- United States (2):
  - The Mind Research Network, Albuquerque, New Mexico
  - The University of New Mexico, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiken, L. S., West, S. G., & Reno, R. R. (1991). Multiple regression: Testing and interpreting interactions. Sage.
- [Background] Allen EA, Erhardt EB, Damaraju E, Gruner W, Segall JM, Silva RF, Havlicek M, Rachakonda S, Fries J, Kalyanam R, Michael AM, Caprihan A, Turner JA, Eichele T, Adelsheim S, Bryan AD, Bustillo J, Clark VP, Feldstein Ewing SW, Filbey F, Ford CC, Hutchison K, Jung RE, Kiehl KA, Kodituwakku P, Komesu YM, Mayer AR, Pearlson GD, Phillips JP, Sadek JR, Stevens M, Teuscher U, Thoma RJ, Calhoun VD. A baseline for the multivariate comparison of resting-state networks. Front Syst Neurosci. 2011 Feb 4;5:2. doi: 10.3389/fnsys.2011.00002. eCollection 2011. PMID 21442040
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Babor, T., Higgins-Biddle, J. C., Saunders, J. B., & Monteiro, M. G. (2001). AUDIT: The Alcohol Use Disorders Identification Test: Guidelines for use in primary care, Second edition. Department of Mental Health and Substance Dependence, World Health Organization.
- [Background] Bechara A, Damasio H. Decision-making and addiction (part I): impaired activation of somatic states in substance dependent individuals when pondering decisions with negative future consequences. Neuropsychologia. 2002;40(10):1675-89. doi: 10.1016/s0028-3932(02)00015-5. PMID 11992656
- [Background] Bechara A, Dolan S, Hindes A. Decision-making and addiction (part II): myopia for the future or hypersensitivity to reward? Neuropsychologia. 2002;40(10):1690-705. doi: 10.1016/s0028-3932(02)00016-7. PMID 11992657
- [Background] Bell AJ, Sejnowski TJ. An information-maximization approach to blind separation and blind deconvolution. Neural Comput. 1995 Nov;7(6):1129-59. doi: 10.1162/neco.1995.7.6.1129. PMID 7584893
- [Background] Bowen S, Chawla N, Collins SE, Witkiewitz K, Hsu S, Grow J, Clifasefi S, Garner M, Douglass A, Larimer ME, Marlatt A. Mindfulness-based relapse prevention for substance use disorders: a pilot efficacy trial. Subst Abus. 2009 Oct-Dec;30(4):295-305. doi: 10.1080/08897070903250084. PMID 19904665
- [Background] Bowen S, Witkiewitz K, Clifasefi SL, Grow J, Chawla N, Hsu SH, Carroll HA, Harrop E, Collins SE, Lustyk MK, Larimer ME. Relative efficacy of mindfulness-based relapse prevention, standard relapse prevention, and treatment as usual for substance use disorders: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):547-56. doi: 10.1001/jamapsychiatry.2013.4546. PMID 24647726
- [Background] Brewer JA, Bowen S, Smith JT, Marlatt GA, Potenza MN. Mindfulness-based treatments for co-occurring depression and substance use disorders: what can we learn from the brain? Addiction. 2010 Oct;105(10):1698-706. doi: 10.1111/j.1360-0443.2009.02890.x. PMID 20331548
- [Background] Calhoun VD, Adali T. Multisubject independent component analysis of fMRI: a decade of intrinsic networks, default mode, and neurodiagnostic discovery. IEEE Rev Biomed Eng. 2012;5:60-73. doi: 10.1109/RBME.2012.2211076. PMID 23231989
- [Background] Calhoun VD, Adali T, Pearlson GD, Pekar JJ. A method for making group inferences from functional MRI data using independent component analysis. Hum Brain Mapp. 2001 Nov;14(3):140-51. doi: 10.1002/hbm.1048. PMID 11559959
- [Background] Cardenas VA, Studholme C, Gazdzinski S, Durazzo TC, Meyerhoff DJ. Deformation-based morphometry of brain changes in alcohol dependence and abstinence. Neuroimage. 2007 Feb 1;34(3):879-87. doi: 10.1016/j.neuroimage.2006.10.015. Epub 2006 Nov 28. PMID 17127079
- [Background] Charlet K, Beck A, Jorde A, Wimmer L, Vollstadt-Klein S, Gallinat J, Walter H, Kiefer F, Heinz A. Increased neural activity during high working memory load predicts low relapse risk in alcohol dependence. Addict Biol. 2014 May;19(3):402-14. doi: 10.1111/adb.12103. Epub 2013 Oct 22. PMID 24147643
- [Background] Charlet K, Schlagenhauf F, Richter A, Naundorf K, Dornhof L, Weinfurtner CE, Konig F, Walaszek B, Schubert F, Muller CA, Gutwinski S, Seissinger A, Schmitz L, Walter H, Beck A, Gallinat J, Kiefer F, Heinz A. Neural activation during processing of aversive faces predicts treatment outcome in alcoholism. Addict Biol. 2014 May;19(3):439-51. doi: 10.1111/adb.12045. Epub 2013 Mar 7. PMID 23469861
- [Background] Claus ED, Ewing SW, Filbey FM, Sabbineni A, Hutchison KE. Identifying neurobiological phenotypes associated with alcohol use disorder severity. Neuropsychopharmacology. 2011 Sep;36(10):2086-96. doi: 10.1038/npp.2011.99. Epub 2011 Jun 15. PMID 21677649
- [Background] Claus ED, Feldstein Ewing SW, Filbey FM, Hutchison KE. Behavioral control in alcohol use disorders: relationships with severity. J Stud Alcohol Drugs. 2013 Jan;74(1):141-51. doi: 10.15288/jsad.2013.74.141. PMID 23200160
- [Background] Claus ED, Hutchison KE. Neural mechanisms of risk taking and relationships with hazardous drinking. Alcohol Clin Exp Res. 2012 Jun;36(6):932-40. doi: 10.1111/j.1530-0277.2011.01694.x. Epub 2012 Feb 6. PMID 22309791
- [Background] Claus ED, Kiehl KA, Hutchison KE. Neural and behavioral mechanisms of impulsive choice in alcohol use disorder. Alcohol Clin Exp Res. 2011 Jul;35(7):1209-19. doi: 10.1111/j.1530-0277.2011.01455.x. Epub 2011 Apr 19. PMID 21676001
- [Background] Claus, E.D., Littlewood, R.A., Feldstein Ewing, S.W., Aranella, P., Bogenschutz, M.P., Hutchison, K.E. (unpublished). BOLD response as a potential biomarker predicting treatment response to olanzapine in alcohol dependence.
- [Background] Conigrave KM, Degenhardt LJ, Whitfield JB, Saunders JB, Helander A, Tabakoff B; WHO/ISBRA Study Group. CDT, GGT, and AST as markers of alcohol use: the WHO/ISBRA collaborative project. Alcohol Clin Exp Res. 2002 Mar;26(3):332-9. PMID 11923585
- [Background] DeVito EE, Worhunsky PD, Carroll KM, Rounsaville BJ, Kober H, Potenza MN. A preliminary study of the neural effects of behavioral therapy for substance use disorders. Drug Alcohol Depend. 2012 May 1;122(3):228-35. doi: 10.1016/j.drugalcdep.2011.10.002. Epub 2011 Oct 29. PMID 22041256
- [Background] Durazzo TC, Gazdzinski S, Mon A, Meyerhoff DJ. Cortical perfusion in alcohol-dependent individuals during short-term abstinence: relationships to resumption of hazardous drinking after treatment. Alcohol. 2010 May;44(3):201-10. doi: 10.1016/j.alcohol.2010.03.003. PMID 20682188
- [Background] Eckardt MJ, Stapleton JM, Rawlings RR, Davis EZ, Grodin DM. Neuropsychological functioning in detoxified alcoholics between 18 and 35 years of age. Am J Psychiatry. 1995 Jan;152(1):53-9. doi: 10.1176/ajp.152.1.53. PMID 7802120
- [Background] Elwafi HM, Witkiewitz K, Mallik S, Thornhill TA 4th, Brewer JA. Mindfulness training for smoking cessation: moderation of the relationship between craving and cigarette use. Drug Alcohol Depend. 2013 Jun 1;130(1-3):222-9. doi: 10.1016/j.drugalcdep.2012.11.015. Epub 2012 Dec 21. PMID 23265088
- [Background] Epstein, E. E. & McCrady, B. S. (2009a). A cognitive-behavioral treatment program for overcoming alcohol use problems: Therapist guide. New York: Oxford University Press.
- [Background] Epstein, E. E. & McCrady, B. S. (2009b). A cognitive-behavioral treatment program for overcoming alcohol use problems: Client workbook. New York: Oxford University Press.
- [Background] Erhardt EB, Rachakonda S, Bedrick EJ, Allen EA, Adali T, Calhoun VD. Comparison of multi-subject ICA methods for analysis of fMRI data. Hum Brain Mapp. 2011 Dec;32(12):2075-95. doi: 10.1002/hbm.21170. Epub 2010 Dec 15. PMID 21162045
- [Background] Filbey FM, Claus E, Audette AR, Niculescu M, Banich MT, Tanabe J, Du YP, Hutchison KE. Exposure to the taste of alcohol elicits activation of the mesocorticolimbic neurocircuitry. Neuropsychopharmacology. 2008 May;33(6):1391-401. doi: 10.1038/sj.npp.1301513. Epub 2007 Jul 25. PMID 17653109
- [Background] Filbey FM, Ray L, Smolen A, Claus ED, Audette A, Hutchison KE. Differential neural response to alcohol priming and alcohol taste cues is associated with DRD4 VNTR and OPRM1 genotypes. Alcohol Clin Exp Res. 2008 Jul;32(7):1113-23. doi: 10.1111/j.1530-0277.2008.00692.x. PMID 18540916
- [Background] Finney, J. W., Moos, R. H., & Timko, C. (2013). The course of treated and untreated substance use disorders: Remission and resolution, relapse and mortality. In: B. S. McCrady & E. e. Epstein (Eds.), Addiction: A comprehensive guidebook, 2nd edition (pp. 108-134). NY: Oxford University Press.
- [Background] First, M. B., William, J. B. W., Karg, R. S., Spitzer, R. L. (2015). User's Guide for the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV). Arlington, VA: American Psychiatric Association.
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Friston, K. J., Ashburner, J., Frith, C. D., Poline, J. B., & Frackowiak, R. S. J. (1995). Spatial registration and normalization of images. Human Brain Mapping, 3, 165-189.
- [Background] Friston, K. J., Holmes, A. P., Worsley, K. J., Poline, J. P., Frith, C. D., & Frackowiak, R. S.J. (1995). Statistical parametric maps in functional imaging: a general linear approach. Human Brain Mapping, 2, 189-210.
- [Background] Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. Psychol Sci. 2007 Mar;18(3):233-9. doi: 10.1111/j.1467-9280.2007.01882.x. PMID 17444920
- [Background] Garland EL, Gaylord SA, Boettiger CA, Howard MO. Mindfulness training modifies cognitive, affective, and physiological mechanisms implicated in alcohol dependence: results of a randomized controlled pilot trial. J Psychoactive Drugs. 2010 Jun;42(2):177-92. doi: 10.1080/02791072.2010.10400690. PMID 20648913
- [Background] Gazdzinski S, Durazzo TC, Studholme C, Song E, Banys P, Meyerhoff DJ. Quantitative brain MRI in alcohol dependence: preliminary evidence for effects of concurrent chronic cigarette smoking on regional brain volumes. Alcohol Clin Exp Res. 2005 Aug;29(8):1484-95. doi: 10.1097/01.alc.0000175018.72488.61. PMID 16131857
- [Background] Grant I, Adams K, Reed R. Normal neuropsychological abilities of alcoholic men in their late thirties. Am J Psychiatry. 1979 Oct;136(10):1263-9. doi: 10.1176/ajp.136.10.1263. PMID 484720
- [Background] Grant BF, Goldstein RB, Saha TD, Chou SP, Jung J, Zhang H, Pickering RP, Ruan WJ, Smith SM, Huang B, Hasin DS. Epidemiology of DSM-5 Alcohol Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions III. JAMA Psychiatry. 2015 Aug;72(8):757-66. doi: 10.1001/jamapsychiatry.2015.0584. PMID 26039070
- [Background] Herault, J., & Jutten, C. (1986). Space or time adaptive signal processing by neural network models. American Institute for Physics Conference Proceedings, 151, 206
- [Background] Heinz A, Wrase J, Kahnt T, Beck A, Bromand Z, Grusser SM, Kienast T, Smolka MN, Flor H, Mann K. Brain activation elicited by affectively positive stimuli is associated with a lower risk of relapse in detoxified alcoholic subjects. Alcohol Clin Exp Res. 2007 Jul;31(7):1138-47. doi: 10.1111/j.1530-0277.2007.00406.x. Epub 2007 May 4. PMID 17488322
- [Background] Jafri MJ, Pearlson GD, Stevens M, Calhoun VD. A method for functional network connectivity among spatially independent resting-state components in schizophrenia. Neuroimage. 2008 Feb 15;39(4):1666-81. doi: 10.1016/j.neuroimage.2007.11.001. Epub 2007 Nov 13. PMID 18082428
- [Background] Jang DP, Namkoong K, Kim JJ, Park S, Kim IY, Kim SI, Kim YB, Cho ZH, Lee E. The relationship between brain morphometry and neuropsychological performance in alcohol dependence. Neurosci Lett. 2007 Nov 20;428(1):21-6. doi: 10.1016/j.neulet.2007.09.047. Epub 2007 Sep 29. PMID 17951002
- [Background] Jutten, C., & Herault, J. (1991). Blind separation of sources, part I: An adaptive algorithm based on neuromimetic architecture. Signal Processing, 24, 1-10.
- [Background] Kareken DA, Claus ED, Sabri M, Dzemidzic M, Kosobud AE, Radnovich AJ, Hector D, Ramchandani VA, O'Connor SJ, Lowe M, Li TK. Alcohol-related olfactory cues activate the nucleus accumbens and ventral tegmental area in high-risk drinkers: preliminary findings. Alcohol Clin Exp Res. 2004 Apr;28(4):550-7. doi: 10.1097/01.alc.0000122764.60626.af. PMID 15100605
- [Background] Kazdin AE, Nock MK. Delineating mechanisms of change in child and adolescent therapy: methodological issues and research recommendations. J Child Psychol Psychiatry. 2003 Nov;44(8):1116-29. doi: 10.1111/1469-7610.00195. PMID 14626454
- [Background] Kiluk BD, Nich C, Babuscio T, Carroll KM. Quality versus quantity: acquisition of coping skills following computerized cognitive-behavioral therapy for substance use disorders. Addiction. 2010 Dec;105(12):2120-7. doi: 10.1111/j.1360-0443.2010.03076.x. Epub 2010 Sep 20. PMID 20854334
- [Background] Kirby KN, Petry NM, Bickel WK. Heroin addicts have higher discount rates for delayed rewards than non-drug-using controls. J Exp Psychol Gen. 1999 Mar;128(1):78-87. doi: 10.1037//0096-3445.128.1.78. PMID 10100392
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Kober H, Mende-Siedlecki P, Kross EF, Weber J, Mischel W, Hart CL, Ochsner KN. Prefrontal-striatal pathway underlies cognitive regulation of craving. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14811-6. doi: 10.1073/pnas.1007779107. Epub 2010 Aug 2. PMID 20679212
- [Background] Koob, G. F. (2013). Neuroscience of addiction. In: B. S. McCrady & E. E. Epstein (Eds.), Addiction: A comprehensive guidebook, 2nd edition (pp. 17-354). NY: Oxford University Press.
- [Background] Koob G, Kreek MJ. Stress, dysregulation of drug reward pathways, and the transition to drug dependence. Am J Psychiatry. 2007 Aug;164(8):1149-59. doi: 10.1176/appi.ajp.2007.05030503. PMID 17671276
- [Background] Lang, P. J., Bradley, M. M., & Cuthbert, B. N. (1997). International affective picture system (IAPS): Technical manual and affective ratings. NIMH Center for the Study of Emotion and Attention, 39-58.
- [Background] Li CS, Luo X, Yan P, Bergquist K, Sinha R. Altered impulse control in alcohol dependence: neural measures of stop signal performance. Alcohol Clin Exp Res. 2009 Apr;33(4):740-50. doi: 10.1111/j.1530-0277.2008.00891.x. Epub 2009 Jan 21. PMID 19170662
- [Background] Loree AM, Lundahl LH, Ledgerwood DM. Impulsivity as a predictor of treatment outcome in substance use disorders: review and synthesis. Drug Alcohol Rev. 2015 Mar;34(2):119-34. doi: 10.1111/dar.12132. Epub 2014 Mar 31. PMID 24684591
- [Background] MacKillop J, Miranda R Jr, Monti PM, Ray LA, Murphy JG, Rohsenow DJ, McGeary JE, Swift RM, Tidey JW, Gwaltney CJ. Alcohol demand, delayed reward discounting, and craving in relation to drinking and alcohol use disorders. J Abnorm Psychol. 2010 Feb;119(1):106-14. doi: 10.1037/a0017513. PMID 20141247
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Magill M, Kiluk BD, McCrady BS, Tonigan JS, Longabaugh R. Active Ingredients of Treatment and Client Mechanisms of Change in Behavioral Treatments for Alcohol Use Disorders: Progress 10 Years Later. Alcohol Clin Exp Res. 2015 Oct;39(10):1852-62. doi: 10.1111/acer.12848. Epub 2015 Sep 7. PMID 26344200
- [Background] Magill M, Longabaugh R. Efficacy combined with specified ingredients: a new direction for empirically supported addiction treatment. Addiction. 2013 May;108(5):874-81. doi: 10.1111/add.12013. Epub 2012 Nov 19. PMID 23072622
- [Background] Maisto SA, Kirouac M, Witkiewitz K. Alcohol use disorder clinical course research: informing clinicians' treatment planning now and in the future. J Stud Alcohol Drugs. 2014 Sep;75(5):799-807. doi: 10.15288/jsad.2014.75.799. PMID 25208198
- [Background] Maisto SA, Roos CR, O'Sickey AJ, Kirouac M, Connors GJ, Tonigan JS, Witkiewitz K. The indirect effect of the therapeutic alliance and alcohol abstinence self-efficacy on alcohol use and alcohol-related problems in Project MATCH. Alcohol Clin Exp Res. 2015 Mar;39(3):504-13. doi: 10.1111/acer.12649. Epub 2015 Feb 19. PMID 25704134
- [Background] McCrady, B. S. (2071). Mechanisms of change and the treatment of alcohol use disorders. In: D. McKay, J. Abramowitz, & E. Storch (Eds.), Mechanisms of syndromes and treatment for psychological problems. NY: Wiley Press.
- [Background] McKeown MJ, Makeig S, Brown GG, Jung TP, Kindermann SS, Bell AJ, Sejnowski TJ. Analysis of fMRI data by blind separation into independent spatial components. Hum Brain Mapp. 1998;6(3):160-88. doi: 10.1002/(SICI)1097-0193(1998)6:3<160::AID-HBM5>3.0.CO;2-1. PMID 9673671
- [Background] Miller, W. R. (1996). Form 90: A structured assessment interview for drinking and related behaviors, test manual. Project MATCH Monograph Series, Vol 5. Bethesda, MD: National Institute of Alcohol Abuse and Alcoholism.
- [Background] Miller, W. R., Mattson, M. E., Arciniega, L. T., Arroyo, J...Zweben, A. (2004). COMBINE behavioral intervention manual. A clinical research guide for therapists treatment people with alcohol abuse and dependence. DHHS Publication No. (NIH) 04-5288. Bethesda, MD: National Institute on Alcohol Abuse and Alcoholism.
- [Background] Miller, W. R. & Rollnick, S. (2013). Motivational interviewing: Helping people change, 3rd edition. NY: Guilford Press.
- [Background] Miller, W.R., Tonigan, J.S. & Longabaugh, R. (1995). The Drinker Inventory of Consequences (DrInC): An instrument for assessing adverse consequences of alcohol abuse. Project MATCH Monograph Series, Vol. 4. DHHS Publication No. 95-3911. Rockville MD: NIAAA.
- [Background] Monnig MA, Tonigan JS, Yeo RA, Thoma RJ, McCrady BS. White matter volume in alcohol use disorders: a meta-analysis. Addict Biol. 2013 May;18(3):581-92. doi: 10.1111/j.1369-1600.2012.00441.x. Epub 2012 Mar 28. PMID 22458455
- [Background] Myrick H, Anton RF, Li X, Henderson S, Randall PK, Voronin K. Effect of naltrexone and ondansetron on alcohol cue-induced activation of the ventral striatum in alcohol-dependent people. Arch Gen Psychiatry. 2008 Apr;65(4):466-75. doi: 10.1001/archpsyc.65.4.466. PMID 18391135
- [Background] Naqvi NH, Morgenstern J. Cognitive Neuroscience Approaches to Understanding Behavior Change in Alcohol Use Disorder Treatments. Alcohol Res. 2015;37(1):29-38. doi: 10.35946/arcr.v37.1.03. PMID 26259087
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Papachristou H, Nederkoorn C, Giesen JC, Jansen A. Cue reactivity during treatment, and not impulsivity, predicts an initial lapse after treatment in alcohol use disorders. Addict Behav. 2014 Mar;39(3):737-9. doi: 10.1016/j.addbeh.2013.11.027. Epub 2013 Dec 11. PMID 24368002
- [Background] Rassen JA, Shelat AA, Franklin JM, Glynn RJ, Solomon DH, Schneeweiss S. Matching by propensity score in cohort studies with three treatment groups. Epidemiology. 2013 May;24(3):401-9. doi: 10.1097/EDE.0b013e318289dedf. PMID 23532053
- [Background] Roos CR, Witkiewitz K. Adding tools to the toolbox: The role of coping repertoire in alcohol treatment. J Consult Clin Psychol. 2016 Jul;84(7):599-611. doi: 10.1037/ccp0000102. Epub 2016 Apr 7. PMID 27054825
- [Background] Rosenbloom M, Sullivan EV, Pfefferbaum A. Using magnetic resonance imaging and diffusion tensor imaging to assess brain damage in alcoholics. Alcohol Res Health. 2003;27(2):146-52. PMID 15303625
- [Background] Rupp CI, Beck JK, Heinz A, Kemmler G, Manz S, Tempel K, Fleischhacker WW. Impulsivity and Alcohol Dependence Treatment Completion: Is There a Neurocognitive Risk Factor at Treatment Entry? Alcohol Clin Exp Res. 2016 Jan;40(1):152-60. doi: 10.1111/acer.12924. Epub 2015 Dec 19. PMID 26683585
- [Background] Sacks JJ, Gonzales KR, Bouchery EE, Tomedi LE, Brewer RD. 2010 National and State Costs of Excessive Alcohol Consumption. Am J Prev Med. 2015 Nov;49(5):e73-e79. doi: 10.1016/j.amepre.2015.05.031. Epub 2015 Oct 1. PMID 26477807
- [Background] Salsman JM, Butt Z, Pilkonis PA, Cyranowski JM, Zill N, Hendrie HC, Kupst MJ, Kelly MA, Bode RK, Choi SW, Lai JS, Griffith JW, Stoney CM, Brouwers P, Knox SS, Cella D. Emotion assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S76-86. doi: 10.1212/WNL.0b013e3182872e11. PMID 23479549
- [Background] Schacht JP, Anton RF, Myrick H. Functional neuroimaging studies of alcohol cue reactivity: a quantitative meta-analysis and systematic review. Addict Biol. 2013 Jan;18(1):121-33. doi: 10.1111/j.1369-1600.2012.00464.x. Epub 2012 May 10. PMID 22574861
- [Background] Schacht JP, Randall PK, Waid LR, Baros AM, Latham PK, Wright TM, Myrick H, Anton RF. Neurocognitive performance, alcohol withdrawal, and effects of a combination of flumazenil and gabapentin in alcohol dependence. Alcohol Clin Exp Res. 2011 Nov;35(11):2030-8. doi: 10.1111/j.1530-0277.2011.01554.x. Epub 2011 Jun 1. PMID 21631542
- [Background] Sebastian A, Baldermann C, Feige B, Katzev M, Scheller E, Hellwig B, Lieb K, Weiller C, Tuscher O, Kloppel S. Differential effects of age on subcomponents of response inhibition. Neurobiol Aging. 2013 Sep;34(9):2183-93. doi: 10.1016/j.neurobiolaging.2013.03.013. Epub 2013 Apr 13. PMID 23591131
- [Background] Seo S, Mohr J, Beck A, Wustenberg T, Heinz A, Obermayer K. Predicting the future relapse of alcohol-dependent patients from structural and functional brain images. Addict Biol. 2015 Nov;20(6):1042-55. doi: 10.1111/adb.12302. Epub 2015 Oct 4. PMID 26435383
- [Background] Silveri MM. Adolescent brain development and underage drinking in the United States: identifying risks of alcohol use in college populations. Harv Rev Psychiatry. 2012 Jul-Aug;20(4):189-200. doi: 10.3109/10673229.2012.714642. PMID 22894728
- [Background] Skinner HA. The drug abuse screening test. Addict Behav. 1982;7(4):363-71. doi: 10.1016/0306-4603(82)90005-3. PMID 7183189
- [Background] Spreng RN, Wojtowicz M, Grady CL. Reliable differences in brain activity between young and old adults: a quantitative meta-analysis across multiple cognitive domains. Neurosci Biobehav Rev. 2010 Jul;34(8):1178-94. doi: 10.1016/j.neubiorev.2010.01.009. Epub 2010 Jan 28. PMID 20109489
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Thayer RE, Hagerty SL, Sabbineni A, Claus ED, Hutchison KE, Weiland BJ. Negative and interactive effects of sex, aging, and alcohol abuse on gray matter morphometry. Hum Brain Mapp. 2016 Jun;37(6):2276-92. doi: 10.1002/hbm.23172. Epub 2016 Mar 7. PMID 26947584
- [Background] Tofighi D, Kelley K. Assessing Omitted Confounder Bias in Multilevel Mediation Models. Multivariate Behav Res. 2016;51(1):86-105. doi: 10.1080/00273171.2015.1105736. PMID 26881959
- [Background] Tofighi D, MacKinnon DP. RMediation: an R package for mediation analysis confidence intervals. Behav Res Methods. 2011 Sep;43(3):692-700. doi: 10.3758/s13428-011-0076-x. PMID 21487904
- [Background] Vollstadt-Klein S, Loeber S, Kirsch M, Bach P, Richter A, Buhler M, von der Goltz C, Hermann D, Mann K, Kiefer F. Effects of cue-exposure treatment on neural cue reactivity in alcohol dependence: a randomized trial. Biol Psychiatry. 2011 Jun 1;69(11):1060-6. doi: 10.1016/j.biopsych.2010.12.016. Epub 2011 Feb 3. PMID 21292243
- [Background] Vollstadt-Klein S, Wichert S, Rabinstein J, Buhler M, Klein O, Ende G, Hermann D, Mann K. Initial, habitual and compulsive alcohol use is characterized by a shift of cue processing from ventral to dorsal striatum. Addiction. 2010 Oct;105(10):1741-9. doi: 10.1111/j.1360-0443.2010.03022.x. PMID 20670348
- [Background] Wechsler, D. (1999). Abbreviated Scale of Intelligence (WASI). San Antonio, Tx.: Harcourt.
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Westbrook C, Creswell JD, Tabibnia G, Julson E, Kober H, Tindle HA. Mindful attention reduces neural and self-reported cue-induced craving in smokers. Soc Cogn Affect Neurosci. 2013 Jan;8(1):73-84. doi: 10.1093/scan/nsr076. Epub 2011 Nov 22. PMID 22114078
- [Background] Whiteside, S. P., Lynam, D. R., Miller, J. D., & Reynolds, S. K. (2005). Validation of the UPPS impulsive behaviour scale: a four-factor model of impulsivity. European Journal of Personality, 19(7), 559-574.
- [Background] Witkiewitz K. Predictors of heavy drinking during and following treatment. Psychol Addict Behav. 2011 Sep;25(3):426-38. doi: 10.1037/a0022889. PMID 21480681
- [Background] Witkiewitz K, Bowen S. Depression, craving, and substance use following a randomized trial of mindfulness-based relapse prevention. J Consult Clin Psychol. 2010 Jun;78(3):362-374. doi: 10.1037/a0019172. PMID 20515211
- [Background] Witkiewitz K, Bowen S, Douglas H, Hsu SH. Mindfulness-based relapse prevention for substance craving. Addict Behav. 2013 Feb;38(2):1563-1571. doi: 10.1016/j.addbeh.2012.04.001. Epub 2012 Apr 6. PMID 22534451
- [Background] Witkiewitz K, Dearing RL, Maisto SA. Alcohol use trajectories among non-treatment-seeking heavy drinkers. J Stud Alcohol Drugs. 2014 May;75(3):415-22. doi: 10.15288/jsad.2014.75.415. PMID 24766753
- [Background] Witkiewitz K, Donovan DM, Hartzler B. Drink refusal training as part of a combined behavioral intervention: effectiveness and mechanisms of change. J Consult Clin Psychol. 2012 Jun;80(3):440-9. doi: 10.1037/a0026996. Epub 2012 Jan 30. PMID 22289131
- [Background] Witkiewitz K, Maisto SA, Donovan DM. A comparison of methods for estimating change in drinking following alcohol treatment. Alcohol Clin Exp Res. 2010 Dec;34(12):2116-25. doi: 10.1111/j.1530-0277.2010.01308.x. Epub 2010 Sep 22. PMID 20860611
- [Background] Witkiewitz K, Marlatt GA. Relapse prevention for alcohol and drug problems: that was Zen, this is Tao. Am Psychol. 2004 May-Jun;59(4):224-35. doi: 10.1037/0003-066X.59.4.224. PMID 15149263
- [Background] Witkiewitz K, Villarroel NA. Dynamic association between negative affect and alcohol lapses following alcohol treatment. J Consult Clin Psychol. 2009 Aug;77(4):633-44. doi: 10.1037/a0015647. PMID 19634957
- [Background] Worhunsky PD, Stevens MC, Carroll KM, Rounsaville BJ, Calhoun VD, Pearlson GD, Potenza MN. Functional brain networks associated with cognitive control, cocaine dependence, and treatment outcome. Psychol Addict Behav. 2013 Jun;27(2):477-88. doi: 10.1037/a0029092. Epub 2012 Jul 9. PMID 22775772